CLINICAL TRIAL: NCT02699073
Title: Evaluation of Treatment Response With CHOI and RECIST Criteria and CT Texture Analysis in Patients With Metastatic Colorectal Cancer Treated With Regorafenib. A GERCOR Phase II Study
Brief Title: Evaluation of Treatment Response With CHOI and RECIST Criteria and CT Texture Analysis in Patients With Metastatic Colorectal Cancer Treated With Regorafenib
Acronym: TEXCAN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEXCAN C15-2
Record Dates: First submitted 2016-02-23; First posted 2016-03-04 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer; metastatic; regorafenib; CHOI criteria; RECIST criteria
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — regorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Regorafenib (Experimental): dose of regorafenib : 160mg once daily
  Interventions: Drug: regorafenib

INTERVENTIONS:
Drug: regorafenib — 160mg once daily during 3 weeks followed by 1 week off therapy.
  Regorafenib will be taken until disease progression according to the CHOI and RECIST1.1 criteria, death or inacceptable toxicity.

SUMMARY:
The purpose of the study is to evaluate the performance of various tumor response criteria (Choi and RECIST1.1 criteria) in the assessment of regorafenib activity.

Moreover, an assessment of the tumor heterogeneity will be made using computed tomographic texture analysis (CTTA)

DETAILED DESCRIPTION:
This is a phase II study in patients with metastatic colorectal cancer treated by regorafenib.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent.
2. Patients with histologically proven metastatic colorectal cancer
3. Patients previously treated with, or who are not considered candidates for available therapies, i.e., fluoropyrimidine-based chemotherapy, anti-VEGF therapy and anti-EGFR therapy (if patients were RAS wild-type).
4. ECOG PS = 0 or 1
5. Aged 18-years or older
6. Life expectancy of at least 3 months
7. Adequate renal, bone marrow, liver and pancreatic functions:

   * Estimated creatinine clearance ≥ 30 mL/min as calculated using the Cockcroft-Gault equation
   * Platelet count ≥ 100.000/mm3; hemoglobin ≥ 9 g/dL; absolute neutrophil count ≥ 1500/mm3. Transfusion to meet the inclusion criteria will not be allowed
   * Total bilirubin ≤ 1.5 the upper limit of normal value (ULN); alanine aminotransferase (ALAT) and aspartame aminotransferase (ASAT) ≤ 3.0 x ULN (≤ 5.0 x ULN for patients with liver involvement of their cancer); alkaline phosphatase (ALP) ≤ 2.5 x ULN (≤ 5.0 x ULN for patients with liver involvement of their cancer and/or have bone metastases)
8. International normalized ratio (INR) ≤ 1.5 x ULN and partial thromboplastin time (PTT) or activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless receiving treatment with therapeutic anticoagulation. Patients being treated with anticoagulant, e.g., heparin, will be allowed to participate provided no prior evidence of an underlying abnormality in these parameters exists. Close monitoring of at least weekly evaluation will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care
9. At least one target lesion on CT scan
10. No contraindication to Iodine contrast media injection during CT.
11. For women of childbearing potential, blood or urine pregnancy test performed a maximum of 7 days before start of study treatment and negative result documented before start of study treatment
12. When applicable, i.e., women of childbearing potential having sexual activity, men having sexual activity, must agree to use an adequate contraception before entering the study, until at least 8 weeks after the last study drug administration
13. Registration in a national health care system (CMU included).

Exclusion Criteria:

1. Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before inclusion in the trial ; planned surgical procedure within the first month of treatment or any procedure that might change the timing of regorafenib administration during the first month of treatment
2. Patients under judicial protection (curatorship, tutorship) and/or deprived of freedom
3. Major surgical procedure, open biopsy or significant traumatic injury within 28 days before start of study medication
4. Pregnancy or breastfeeding
5. Congestive heart failure ≥ New York Heart Association (NYHA) class 2
6. Unstable angina (angina symptoms at rest), new-onset angina (begun within the last 3 months)
7. Myocardial infarction less than 6 months before the start of study medication
8. Cardiac arrhythmias requiring anti-arrhythmic therapy (beta-blockers or digoxin are permitted)
9. Uncontrolled hypertension (systolic blood pressure >140 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
10. Arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within 6 months before the start of study medication (except for adequately treated catheter-related venous thrombosis occurring more than one month before the start of study medication
11. Pleural effusion or ascites that causes respiratory compromise (≥ CTCAE grade 2, NCI-CTCAE v 4.0 dyspnea)
12. Ongoing infection >grade 2, NCI- CTCAE v 4.0
13. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to inclusion, except for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors (Ta [non-invasive tumor], Tis [carcinoma in situ] and T1 [tumor invades lamina propria])
14. Known history of human immunodeficiency virus (HIV) infection
15. Active hepatitis B or C or chronic hepatitis B or C requiring treatment with antiviral therapy
16. Patients with seizure disorder requiring medication
17. History of organ allograft
18. Patients with evidence or history of any bleeding diathesis, irrespective of severity
19. Any hemorrhage or bleeding event ≥ Grade 3, NCI-CTCAE v 4.0 within 4 weeks prior to the start of study medication
20. Non-healing wound, non-healing ulcer or non-healing bone fracture
21. Dehydration grade ≥1, NCI-CTCAE v 4.0
22. Known hypersensitivity to the study drug, study drug classes or excipient in the formulation
23. Interstitial lung disease with ongoing signs or symptoms at the time of inclusion
24. Persistent proteinuria >3.5 g/24 hour measured by urine protein-creatinine ratio from a random urine sample (≥ Grade 3, NCI-CTCAE v 4.0)
25. Patients unable to swallow oral medication
26. Any malabsorption condition
27. Unresolved toxicity higher than Grade 1, NCI-CTCAE v 4.0, attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neuropathy
28. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy, and hormonal therapy during this trial or within 3 weeks
29. Treatment with any other investigational medicinal product within 28 days prior to study entry
30. Chronic treatment potentially interacting with the study medication, i.e. strong CYP3A4 inducers/inhibitors, strong UGT1A9 inhibitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2018-07-09 (Actual)

PRIMARY OUTCOMES:
Tumor response rate at 2 months according Choi Criteria | 2 months after the beginning of treatment

SECONDARY OUTCOMES:
Tumor response rate at 1 and 2 months according to RECIST1.1 | At 1 month and 2 months after the beginning of treatment
Tumor response rate at 1 month according to Choi criteria | At 1 month after the beginning of treatment
Best overall response rate (BOR) according to Choi criteria and to RECIST 1.1 | BOR is the best response recorded from the strat of treatment until treatment failure up to 36 months
Disease control rate (DCR) | DCR is the proportion of patient with tumor response (CR or RP) or tumor stabilization as best response from the inclusion until treatment failure, up to 36 months
Overall Survival (OS) | Assessed from the date of study drug start to the date of patient death, due to any cause or to the last date the patient was known to be alive, up to 36 months
Progression free survival (PFS) | PFS is the time from the date of study drug start to the date of progressive disease or death due to any cause, up to 36 months
Specificity of Choi criteria at 1 month in identifying patients with long or short OS (using median OS as cut-off value). | At 1 month after inclusion
Evaluation of tumor heterogeneity with TexRAD software | At baseline and 1 month after inclusion
  Threshold of the CTTA parameters (Skewness, Kurtosis, Entropy, Uniformity) provided by the TexRAD software at baseline and optimal variations of these parameters on the CT performed at one month (compared to baseline).
Serious adverse events( SAE) and adverse event (AE) | Up to 36 months
  assessed by NCI-CTCAE4.0
Identify early prognostic biomarkers of regorafenib | at baseline, Cycle 1 Day 15, cycle 2 Day 15 and end of treatment
Correlation between Baseline cell free DNA and survival outcomes (PFS and OS) | at baseline, Cycle 1 Day 15, cycle 2 Day 15 and end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Thierry ANDRE, MD, Principal Investigator — Hôpital Saint Antoine
Locations (8):
- France (8):
  - CHU Jean Minjoz, Besançon
  - Hôpitlal Henri Mondor, Créteil
  - Institut Hospitalier Franco-Britannique, Levallois-Perret
  - CHRU Claude Huriez, Lille
  - ICM Val D'Aurelle, Montpellier
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Saint Antoine, Paris
  - Insitut Mutualiste Montouris, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rousseau B, Boukerma AK, Henriques J, Cohen R, Lucidarme O, Borg C, Tournigand C, Kim S, Bachet JB, Mazard T, Louvet C, Chibaudel B, Vernerey D, Andre T, Hulin A. Impact of trough concentrations of regorafenib and its major metabolites M-2 and M-5 on overall survival of chemorefractory metastatic colorectal cancer patients: Results from a multicentre GERCOR TEXCAN phase II study. Eur J Cancer. 2022 Jun;168:99-107. doi: 10.1016/j.ejca.2022.03.009. Epub 2022 Apr 27. PMID 35489233
- [Derived] Lucidarme O, Wagner M, Gillard P, Kim S, Bachet JB, Rousseau B, Mazard T, Louvet C, Chibaudel B, Cohen R, Garcia-Larnicol ML, Gobert A, Henriques J, Andre T. RECIST and CHOI criteria in the evaluation of tumor response in patients with metastatic colorectal cancer treated with regorafenib, a prospective multicenter study. Cancer Imaging. 2019 Dec 9;19(1):85. doi: 10.1186/s40644-019-0271-z. PMID 31818317